CLINICAL TRIAL: NCT03697954
Title: Direct Full-stage Implantation of Sacral Neuromodulation
Status: Withdrawn | Type: Observational
Why Stopped: Work has already been published by other groups
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Andrea Staack, MD PhD, Loma Linda University
Other Study IDs: 5180114
Record Dates: First submitted 2018-10-04; First posted 2018-10-05 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Urinary Bladder, Overactive; Urge Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- overactive bladder patients: Female patients with refractory overactive bladder and urge urinary incontinence undergoing direct full stage implantation
  Interventions: Device: full stage implantation of sacral neuromodulation

INTERVENTIONS:
Device: full stage implantation of sacral neuromodulation — full stage implantation of sacral neuromodulation for overactive bladder and urge incontinence

SUMMARY:
The purpose of this investigator-initiated study is to investigate the efficacy and costs of direct full stage sacral neuromodulation in patients with overactive bladder. Patients with refractory OAB and urge urinary incontinence will undergo direct full stage implantation and be followed for a period of 6 months to monitor symptom improvement with voiding diaries and validated questionnaires preoperatively and postoperatively. Therapeutic and adverse outcomes will be evaluated. The use of medical resources and time off of work will be analyzed as well. This will be a descriptive study with no additional arms or randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* Female gender
* Refractory overactive bladder: wet failing treatment with two or more anticholinergic and/or beta-3 agonist agents
* Willing to stop treatment with anticholingeric and/or beta-3 agonist agents during the study period (2 week washout period preoperatively and 6 months postoperative)
* Willing and able to complete study questionnaires, use Medtronic device programmer, return for scheduled follow-up appointments
* Surgical candidate able to hold antiplatelet or anticoagulation prior to surgery
* Health insurance provider that will cover full-stage implantation

Exclusion Criteria:

* Age <18
* Pregnant or planning to become pregnant
* Male gender
* Unable or unwilling to stop anticholingeric and/or beta-3 agonist agents during the study period
* Treatment with botulinum toxin within last 6 months
* Recent surgery for stress urinary incontinence or pelvic organ prolapse within last 6 months
* Severe pelvic organ prolapse
* Post-void residual >150 ml
* Symptomatic or recurrent urinary tract infection
* Neurologic disorders: cerebrovascular accident with neurologic deficits, Parkinson's, multiple sclerosis, spinal cord injury, significant peripheral neuropathy
* Cognitive disorders, e.g. dementia
* Interstitial cystitis or chronic pelvic pain syndrome
* Poorly controlled diabetes mellitus (HbA1c >10%)
* History of bladder malignancy, pelvic radiation, urinary retention requiring catheterization
* Anticipated or known need for MRI at the trunk
* History of or anticipated surgery at the lower back
* Unable to hold antiplatelet or anticoagulation prior to surgery
* Life expectancy <1 year

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Patients with refractory overactive bladder and urge urinary incontinence undergoing direct full stage implantation.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in overactive bladder symptoms | 1 year
  measured using overactive bladder questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University Faculty Medical Offices, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Irwin DE, Kopp ZS, Agatep B, Milsom I, Abrams P. Worldwide prevalence estimates of lower urinary tract symptoms, overactive bladder, urinary incontinence and bladder outlet obstruction. BJU Int. 2011 Oct;108(7):1132-8. doi: 10.1111/j.1464-410X.2010.09993.x. Epub 2011 Jan 13. PMID 21231991
- [Background] Ganz ML, Smalarz AM, Krupski TL, Anger JT, Hu JC, Wittrup-Jensen KU, Pashos CL. Economic costs of overactive bladder in the United States. Urology. 2010 Mar;75(3):526-32, 532.e1-18. doi: 10.1016/j.urology.2009.06.096. Epub 2009 Dec 29. PMID 20035977
- [Background] Coyne KS, Sexton CC, Irwin DE, Kopp ZS, Kelleher CJ, Milsom I. The impact of overactive bladder, incontinence and other lower urinary tract symptoms on quality of life, work productivity, sexuality and emotional well-being in men and women: results from the EPIC study. BJU Int. 2008 Jun;101(11):1388-95. doi: 10.1111/j.1464-410X.2008.07601.x. PMID 18454794
- [Background] Latini JM, Alipour M, Kreder KJ Jr. Efficacy of sacral neuromodulation for symptomatic treatment of refractory urinary urge incontinence. Urology. 2006 Mar;67(3):550-3; discussion 553-4. doi: 10.1016/j.urology.2005.09.066. PMID 16527577
- [Background] Gormley EA, Lightner DJ, Burgio KL, Chai TC, Clemens JQ, Culkin DJ, Das AK, Foster HE Jr, Scarpero HM, Tessier CD, Vasavada SP; American Urological Association; Society of Urodynamics, Female Pelvic Medicine & Urogenital Reconstruction. Diagnosis and treatment of overactive bladder (non-neurogenic) in adults: AUA/SUFU guideline. J Urol. 2012 Dec;188(6 Suppl):2455-63. doi: 10.1016/j.juro.2012.09.079. Epub 2012 Oct 24. PMID 23098785